CLINICAL TRIAL: NCT00239330
Title: An Open-label, Randomised, Multi-centre, Phase IIIb, Parallel Group Study to Compare the Efficacy and Safety of Rosuvastatin and Atorvastatin in Subjects With Type IIa and IIb Hypercholesterolaemia
Brief Title: Direct Statin Comparison of LDL-C Values: an Evaluation of Rosuvastatin Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3560L00011; DISCOVERY
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Hypercholesteremia
Keywords: high blood cholesterol levels
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium; Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor
Drug: Atorvastatin

SUMMARY:
The primary objective of the study is to compare the efficacy of rosuvastatin 10 mg with atorvastatin 10 mg by assessment of the percentage of subjects who reach EAS LDL-C target goals after 12 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, age > 18 years
* Primary hypercholesterolaemia with CV risk > 20% (as defined in European Guidelines ) and/or type II diabetes and/or a history of CHD or other established atherosclerotic disease. Subjects may be lipid-lowering therapy naïve or have been treated for min. 4 weeks with a 'start' dose of any lipid-lowering therapy, which was ineffective.
* Naïve subjects must have completed 12-weeks dietary counselling before this visit.

Exclusion Criteria:

* Known heterozygous or homozygous familial hypercholesterolaemia or known type III hyperlipoproteinaemia (familial dysbetalipoproteinaemia).
* Documented secondary hypercholesterolaemia of any cause other than named in inclusion criteria 3.
* Serious or unstable medical condition
* Statin contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 824
Dates: Start 2003-06; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to compare the efficacy of rosuvastatin 10 mg with atorvastatin 10 mg by assessment of the percentage of subjects who reach EAS LDL-C target goals after 12 weeks of therapy.

SECONDARY OUTCOMES:
To compare the efficacy of rosuvastatin 10 mg with atorvastatin 10 mg by assessment of the percentage of subjects who reach EAS TC treatment goal after 12 weeks of therapy.
To compare the percentage change in LDL-C, TC, HDL-C and TG from pre-dose rosuvastatin 10 mg / atorvastatin 10 mg (week 0) and at 12 weeks. This will be performed separately for the switched and the naïve subjects.
To compare the efficacy of rosuvastatin 10 mg with atorvastatin 10 mg in modifying lipids (Non-HDL-C, TC/HDL-C, LDL-C/ HDL-C, non-HDL-C/HDL-C) at week 12. This will be performed separately for the switched and the naïve subjects.
To compare rosuvastatin 10 mg with atorvastatin 10 mg after 12 & 24 weeks of treatment with respect to the incidence & severity of adverse events & abnormal laboratory values.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Vandenhoven, MD, Study Director — AstraZeneca NV/SA
Locations (26):
- Belgium (26):
  - Research Site, Antwerp
  - Research Site, Arlon
  - Research Site, Assebroek
  - Research Site, Ath
  - Research Site, Aye
  - Research Site, Bastogne
  - Research Site, Baudour
  - Research Site, Borgerhout
  - Research Site, Bornem
  - Research Site, Bouge
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Dendermonde
  - Research Site, Frameries
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Havré
  - Research Site, Kortenberg
  - Research Site, Leuven
  - Research Site, Mol
  - Research Site, Namur
  - Research Site, Ostend
  - Research Site, Roeselare
  - Research Site, Schoten
  - Research Site, Sint-Agatha-Berchem